CLINICAL TRIAL: NCT03610412
Title: Effect of Cinnamomum Cassia as an Enhancer of the Insulin Response of the Insulin-Like Growth Factor-1 and Metabolic Control in Patients With Type 2 Diabetes Mellitus Treated With Metformin Without Glycemic Control
Brief Title: Cinnamomum Cassia Effect on IGF1 and Metabolic Control in Patients With DM2 Without Glycemic Control Metformin Treated
Acronym: CICAFAC1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Sandra Ofelia Hernández González, Medical Research Associate C, Unit in Clinical Epidemiology, Specialities Hospital, Medical Unit of High Specialty; West National Medical Center, Mexican Institute of Social Security., Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2018-1301-031
Record Dates: First submitted 2018-03-23; First posted 2018-08-01 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus Type 2; IGF1; Cinnamomum cassia; Metabolic control; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial, of two parallel groups, double blind, with random assignment and control group.
  Process:
  Visit 1 / Day -7: Period of scrutiny, study information, consent signature, clinical history, anthropometry, baseline laboratory tests.
  Visit 2 / Day 0: Start the intervention period, simple random assignment for study groups, delivery of medication, general recommendations of diet and exercise.
  Visit 3 / Day 30 - Visit 4 / Day 60: Adherence to treatment, taking laboratory tests, evaluation of adverse events, general recommendations of diet and exercise, general recommendations of diet and exercise will be evaluated.
  Final Visit / Day 90 ± 7: Anthropometric measurements will be taken, laboratory tests will be taken, treatment adherence and adverse events will be evaluated, end of the intervention period.
Who Masked: Participant, Investigator
Masking Description: Random assignment of groups and blinding:
  All participants will be submitted to the selection of a sealed envelope which will have a numerical code previously defined by a third party for each intervention group.
  The total number of envelopes required to complete the minimum number of participants (28) will be divided according to sex in two boxes, there will be 14 envelopes for men and 14 envelopes for women, with numerical codes that identify the bottle of intervention treatment that should receive the participant during the intervention period. They will be divided into 7 blinded codes for cinnamomum cassia group and 7 for placebo to complete the size of each subsample. Chance guarantees blinding, neither the participant nor the researcher will know the type of treatment. The database for the blinded statistical analysis will be completed. The blind man will be removed once the statistical analysis has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamomum Cassia (Active Comparator): A group of 14 patients (7 women and 7 men) with DM2 without adequate control, treated with metformin 850mg daily, who will receive 1g of cinnamomum cassia orally every 8 hours, for 90 days.
  Interventions: Other: Cinnamomum Cassia
- Placebo (Placebo Comparator): A group of 14 patients (7 women and 7 men) with DM2 without adequate control, treated with metformin 850mg daily, who will receive 1g of placebo (calcined magnesia) orally every 8 hours, for 90 days.
  Interventions: Other: Placebo (calcined magnesia)

INTERVENTIONS:
Other: Cinnamomum Cassia — The intervention period will be 90 days, unlike other trials with Cinnamomum cassia and the main effect sought is on IGF1 levels, in addition to metabolic control.
  Arms: Cinnamomum Cassia
Other: Placebo (calcined magnesia) — The intervention period will be 90 days, unlike other trials with Cinnamomum cassia and comparison with placebo. The main effect sought is on IGF1 levels, in addition to metabolic control.
  Arms: Placebo

SUMMARY:
Among the multiple treatment options for Diabetes Mellitus Type 2 (DM2), the influence on Insuline like growth factor 1 (IGF1) plays a causal role in diabetes but has shown similarities with insulin, both in its structure and in its function, including a rapid reduction in glucose levels in blood, could improve glycemic control in patients.

Oral administration of 3 g of cinnamomum cassia for 90 days acts as an enhancer of the IGF1 insulin response and on metabolic control (fasting glucose, glycosylated hemoglobin (HbA1c), triglycerides, total cholesterol, high density cholesterol, low density cholesterol, very low density cholesterol, systolic and diastolic blood pressure (TAS and TAD), body weight) in patients with DM2 without glycemic control treated with metformin at doses ≤ 850 mg daily.

DETAILED DESCRIPTION:
Introduction:

DM2 is a chronic disease, considered a public health problem, scenario in which each year increases the number of people affected, has a high prevalence in the investigator's country, 9.4% (ENSANUT 2016), which causes a high morbidity and mortality. Conceptually it is defined as a heterogeneous syndrome originated by the genetic-environmental interaction and characterized by a chronic hyperglycemia, as a consequence of a deficiency in the secretion or action of insulin, which triggers acute complications (ketoacidosis and hyperosmolar coma), microvascular chronicles (retinopathies) and neuropathies) and macrovascular (coronary heart disease, cerebrovascular and peripheral vascular diseases).

Growth hormones such as IGF1 with important biological effects on metabolism have been shown to promote the absorption of glucose in certain peripheral tissues. It has been shown that IGF1 binds to insulin receptors to stimulate the transport of glucose in fat and muscle, inhibiting the production of hepatic glucose by lowering blood glucose while at the same time suppressing insulin secretion, increasing sensitivity to insulin and improves the lipid profile.

For the treatment of DM2 the use of botanical products can improve glucose metabolism by hypoglycemic effect, as well as that of lipids and antioxidant, aqueous extracts of cinnamomum cassia have been shown to enhance glucose uptake and glycogen synthesis in vitro and increase phosphorylation of the insulin receptor with possible effect on IGF1 receptor.

The emergence of other therapies can generate new treatments for patients with DM2, which in turn reduce costs and help improve the quality of life.

Justification:

The prevalence of diabetes and metabolic decontrol is high both in Mexico and in the world and conditions the development of long-term complications. The concentrations of IGF1 in blood are diminished in the patients with diabetes mellitus and by its effects similar to the insulin in the metabolism of the glucose when normalizing this can produce control of the diabetes.

In vitro studies have shown that cinnamomum cassia increases glucose uptake, glycogen synthesis and insulin receptor phosphorylation. In humans it has been confirmed that it increases the levels of glucagon-like peptide 1 (GLP-1), favors the activation of peroxisome proliferator-activated receptor (PPAR-γ and PPAR-α) promoting insulin sensitivity, as well as inhibits hepatic 3-hydroxy 3-methylglutaryl coenzyme A reductase to reduce the synthesis of cholesterol and has a vasodilator effect by activity on the enzyme nitric oxide synthase.

Cinnamomum cassia also has a proposal on the signaling of IGF1 receptors (GRB2), which activated by phosphatidylinositol 3-kinase (PI3K) control the proliferation of IGF1, this IGF1 having reduced levels in patients with diabetes becomes a therapeutic target for improved control metabolic. However, the direct application of IGF1 has as main limitation important collateral effects which has inhibited its use, so it is intended to evaluate the stimulatory effect on IGF1 with cinnamomum cassia considering phytopharmaceutical of good quality and low side effects.

General hypothesis:

Cinnamomum cassia acts as an enhancer of the insulin response of IGF1 and metabolic control in patients with DM2 without glycemic control treated with metformin at low doses.

Goals:

GENERAL To evaluate the effect of cinnamomum cassia as an enhancer of the insulin response of IGF1 on metabolic control in patients with DM2 without glycemic control treated with metformin.

SPECIFIC

To analyze the effect before and after daily oral administration of 850mg of metformin plus 3g of cinnamomum cassia compared to placebo for 90 days on:

* Levels of IGF1.
* Fasting glucose value, HbA1c, triglycerides, total cholesterol, high density cholesterol, low density cholesterol, very low density cholesterol, systolic and diastolic blood pressure, body weight.

SECONDARY

To analyze the effect before and after daily oral administration of 850mg of metformin plus 3g of cinnamomum cassia compared to placebo for 90 days on:

* Insulin sensitivity, body mass index (BMI), waist circumference, % body fat.
* Determine the pharmacological attachment and tolerability of CC and placebo.

Working universe:

Patients with DM2, (men and women with a recent diagnosis, treated with 850 mg of metformin daily, without glycemic control). Residents of Guadalajara and metropolitan area and that for the development of the protocol they will go to the facilities of the National Medical Center of the West, Specialty Hospital.

Sample size:

It was calculated according to the following formula for clinical trials: n= 2 [ (Zα - Z1-β) (δ) / d] 2 Two working groups will be formed at random, which will be integrated as follows: 1) a group of 14 patients (7 women and 7 men) with DM2 without adequate control, treated with metformin 850 mg daily, who will receive 1 g of cinnamomum cassia orally every 8 hours, for 90 days, and 2) a group of 14 patients (7 women and 7 men) with DM2 without adequate control, treated with metformin 850 mg daily, who will receive 1 g of placebo (calcined magnesia ) orally every 8 hours, for 90 days. In this way, the total number of participants required for the study will be, at least, 28 volunteers.

Variables:

Independent variable:

Pharmacological intervention:

* Intervention group: Administration of metformin 850mg daily and cinnamomum cassia 1g orally before each meal, for 90 days.
* Control group: Administration of metformin 850mg daily and of placebo approved 1g (calcined magnesia) orally before each meal, for 90 days.

Dependent variables:

Primary outcome dependent variables:

* Laboratory determinations: IGF1, fasting glucose, HbA1c, lipid profile.
* Clinical determinations: systolic and diastolic blood pressure, body weight.

Dependent secondary outcome variables:

* Laboratory determinations: serum creatinine, liver profile.
* Clinical determinations: Insulin sensitivity, body mass index, waist circumference and percentage of adiposity.

Intervening variables:

* Diet.
* Exercise and physical activity.
* Phase of the menstrual cycle.
* Age.
* Gender.

Clinical procedures:

All the anthropometric and vital signs determinations, as well as the procedures for the interrogation, physical examination and integration of the corresponding clinical history will be carried out by means of universally accepted methods and in accordance with the General Health Law, in its Regulation on the Provision of Medical Care Services.

The history and clinical exploration will be performed at the first visit of the participant in order to establish eligibility to continue in the study. All positive and clinically interesting data will be recorded in the data collection notebook (CRD).

Paraclinical procedures:

During each of the scheduled visits to the research unit it will be necessary to determine a clinical chemistry study, for this purpose it will be essential to collect blood samples and their subsequent processing. For the collection of all blood samples in each of the visits to the research center all participants will be cited at 8:00 am and will be an indispensable requirement in each of the collections of samples that come in a fasting state of 12 hours.

Once the blood sample has been taken, the patient will be given general guidance and recommendations on diet and exercise for a healthy lifestyle. From the 3rd visit the attachment to the treatment will be evaluated, this determination will be made with the following formula, considering as acceptable a value ≥ 80%:

Compliance rate (%) = Total number of capsules you ingested / Total number of capsules you should have ingested = Result multiplied by 100.

Quality control in procedures:

The quality and information management procedures will have the following quality control strategies:

* Review of the database in duplicate.
* Electronic comparison of duplicate database.
* Statistical review of the quality of the information.
* Statistical adjustment of the information.
* Calculation in duplicate of the statistical parameters of quality control.

Data management and analysis:

Database All participants will have a complete clinical record during the development of the study. All the clinical and biochemical data that are submitted to statistical analysis must be registered in the corresponding CRD of each participant. The database will be developed from the CRDs, according to the coding included in said document, in * .xls format of the Microsoft Excel program. Updating and verification of the initial database will be done every time new data is obtained throughout the development of the field work. Once all the participants complete all the visits of the field work phase of the study, a review, verification and final validation of the initial database will be carried out. When the absence of errors in the initial database is verified, it will be converted to the format for analysis under the statistical package SPSS version 21 or higher for Windows.

Statistic analysis:

The most appropriate and reliable statistical procedures for the analysis of the data will be decided based on the result of the normality test. Overall the descriptive statistics used in the presentation of the data will include qualitative measures in frequency and percentage and quantitative measures of central tendency and dispersion (arithmetic mean and standard deviation), when considered appropriate it will also include median, minimum and maximum values or dispersion ranges.

For all cases, the significance will be p ≤ 0.05. All patients receiving at least one dose of intervention treatment will be taken into account in the statistical analysis as part of the intention-to-treat analysis of the eliminated subjects.

Ethical and legal framework:

All the procedures and activities carried out during the development of this clinical trial will be carried out in full compliance with the legal provisions of the General Health Law of the United Mexican States, and in accordance with the ethical principles for pharmacological research on human beings detailed in the latest revision of the Helsinki Declaration and the International Harmonization Conference.

The research protocol will be submitted for approval by the local Research Committee of the Specialties Hospital of the National Medical Center of the West. The study is classified within the General Health Law and its regulations on research in humans as of risk greater than the minimum, since it is a pharmacological study with potential risk; for which it is required to obtain a consent under written information signed at the beginning of the study. The document will be signed in duplicate by the participant, two witnesses from outside the research team and preferably relatives or friends of the participant, and by the principal investigator of the center. One of the duplicates of informed consent will remain with the principal investigator, while the other will be delivered to the study participant.

According to the guidelines of good clinical practice all participants in the study will be identified only by initials and number in the database. The records and laboratory results will be available only to the principal investigators, and with the restrictions of law for the participant.

Conflicts of interest:

There are no conflicts of interest for the conduct of the study. The information obtained from this study will be made available to privileged researchers involved in the development of it.

ELIGIBILITY:
Inclusion Criteria:

* Signature of consent under written information prior to the completion of any procedure in the study.
* Men and women aged 40 to 59 years old, residents of Guadalajara, Jalisco and the metropolitan area.
* Ability to communicate and meet all the requirements of the study.
* BMI less than or equal to 34.9 kg / m2.
* Diagnosis of DM2 according to the ADA:

  * Plasmatic glucose ≥126mg / dl (7.0 mmol / L) in an 8-hour fast.
  * Plasmatic glucose ≥200mg / dl (11.1 mmol / L) at 2 hours after an oral glucose tolerance test.

or HbA1C ≥6.5% (48 mmol / mol).

o Plasmatic glucose ≥200mg / dl (11.1 mmol / L) in a random sample to the patient with classic symptoms of hyperglycemia.

* Evolution of DM2 less than 1 year.
* Be receiving pharmacological treatment with metformin in doses less than or equal to 850mg.
* Stable body weight within 3 months prior to the start of the study, defined as a variability in body weight of less than 10%.
* Eumenorrheic women with mechanical or definitive contraceptive method without hormonal treatment.

Exclusion Criteria:

* Determination of HbA1c less than 6.5%, greater than 10% or fasting glucose greater than 250 mg / dL.
* Serum total cholesterol concentration greater than or equal to 240mg / dl.
* Serum triglyceride concentration greater than or equal to 400mg / dl.
* History of hypersensitivity to study drugs.
* Intake of drugs with known effects on glucose metabolism, lipids, and weight.
* Uncontrolled arterial hypertension, defined as systolic blood pressure values greater than or equal to 140mm / Hg and a diastolic blood pressure greater than or equal to 90mm / Hg.
* History of cardiovascular disease, blood disorders, kidney, pancreatic or thyroid disease.
* Women with suspicion or confirmation of pregnancy
* Women in breastfeeding period.
* History of smoking at any intensity within 12 months prior to the start of the study.
* History of drug abuse or alcoholism.
* Inability to attend or answer the evaluations made in each of the visits.
* Pacemaker bearing, or any other permanent bioelectronic element that can modify the electric bioimpedance reading or be affected by it.

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The sample size will be 28 patients, 14 men and 14 women.
Enrollment: 28 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
The effect of cinnamomum cassia on IGF1 levels. | 90 days
  Changes in the levels of IGF1
The effect of cinnamomum cassia potentiates the insulin response of IGF1 on metabolic control in patients with DM2 without glycemic control treated with metformin. | 90 days
  Changes in the levels of the fasting glucose decrease and glycated hemoglobin
The effect of cinnamomum cassia on metabolic control in patients with DM2 without glycemic control treated with metformin | 90 days
  Changes in the levels of total cholesterol
The effect of cinnamomum cassia on metabolic control | 90 days
  Changes in the levels of tryglicerides
The effect of cinnamomum cassia on blood pressure | 90 days
  Changes in the levels of systolic and diastolic blood pressure
The effect of cinnamomum cassia on body weight | 90 days
  Changes in the body weight

SECONDARY OUTCOMES:
The effect of cinnamomum cassia potentiates the IGF1 insulin response on insulin sensitivity. | 90 days
  Changes in insulin sensitivity.
The effect of cinnamomum cassia potentiates the IGF1 insulin response on BMI. | 90 days
  Changes in body mass index..
The effect of cinnamomum cassia potentiates the IGF1 insulin response on waist circumference. | 90 days
  Changes in waist circumference.
The effect of cinnamomum cassia potentiates the IGF1 insulin response on body fat%. | 90 days
  Changes in body fat percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra O Hernández González, Doctorado, Principal Investigator — Instituto Mexicano del Seguro Social, Unidad de Investigación Biomédica 02
Locations (1):
- Biomedical Unit Research 02, Specialties Hospital, Medical Unit of High Specialty, West National Medical Center, Mexican Social Security Institute., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All data resulting from the clinical investigation, except the personal identification of the subjects (name, address, telephone, etc.)
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication.
Access Criteria: The data can be shared through a request addressed to the principal investigator Dr. Sandra Ofelia Hernández González, basing the reason for what they are requested.

REFERENCES:
- [Background] Sonne DP, Hemmingsen B. Comment on American Diabetes Association. Standards of Medical Care in Diabetes-2017. Diabetes Care 2017;40(Suppl. 1):S1-S135. Diabetes Care. 2017 Jul;40(7):e92-e93. doi: 10.2337/dc17-0299. No abstract available. PMID 28637892
- [Background] Organización Mundial de la Salud. Informe mundial sobre la diabetes. Ginebra, 2016
- [Background] Instituto Nacional de Salud Pública. Encuesta Nacional de Salud y Nutrición de Medio Camino 2016 Informe Final de Resultados. 2016.
- [Background] Asociación Latinoamericana de Diabetes. Consenso de Prediabetes. Documento de Posición de la Asociación Latinoamericana de Diabetes (ALAD) 2016.
- [Background] National Institute for Health and Care Excellence. Preventing type 2 diabetes: risk identification and interventions for individuals at high risk. Public health guideline [PH38] 2012.
- [Background] Bautista Rodríguez LM, Zambrano Plata GE. La calidad de vida percibida en pacientes diabéticos tipo 2. Investigación en Enfermería: Imagen y Desarrollo. 2015;17(1):131-148.
- [Background] Guía de Práctica Clínica. Diagnóstico y tratamiento de la retinopatía diabética, 2015. Guía de Referencia Rápida. Catálogo Maestro de Guías de Práctica Clínica: Actualización 2015, IMSS-171-09
- [Background] Chiarelli F, Trotta D, Verrotti A, Mohn A. Kidney involvement and disease in patients with diabetes. Panminerva Med. 2003 Mar;45(1):23-41. PMID 12682618
- [Background] Najafian B, Alpers CE, Fogo AB. Pathology of human diabetic nephropathy. Contrib Nephrol. 2011;170:36-47. doi: 10.1159/000324942. Epub 2011 Jun 9. PMID 21659756
- [Background] Pedraza L. Diabetic neuropathies: classification and diagnosis. Rev. Med. Clin. Condes 2009; 20(5) 681-686.
- [Background] Julio RA. Galleguillos I. Diabetes and peripheral vascular disease. Rev. Med. Clin. Condes 2009; 20(5) 687-697.
- [Background] Ampudia-Blasco FJ, Navarro J. [Cardiovascular disease in diabetes mellitus]. Med Clin (Barc). 2002 Mar 9;118(8):306-11. doi: 10.1016/s0025-7753(02)72367-1. No abstract available. Spanish. PMID 11888500
- [Background] Arauza A, Ruíz-Franco A. Enfermedad vascular cerebral. Rev Fac Med UNAM 2012; 55 (3): 11-21.
- [Background] Ruiz-Sandoval JL, Leon-Jimenez C, Chiquete-Anaya E, Sosa-Hernandez JL, Espinosa-Casillas CA, Cantu C, Villarreal J, Barinagarrementeria F, Ruiz-Sandoval JL, Arauz A, Leyva A, Murillo L, Alegria MA, Merino J, Romano J, Gonzalez-Vargas O; Asociacion Mexicana de Enfermedad Vascular Cerebral. [Lifestye and primary and secondary prevention for cerebrovascular disease]. Rev Invest Clin. 2010 Mar-Apr;62(2):181-91. No abstract available. Spanish. PMID 20597398
- [Background] Cervantes-Villagrana RD, Presno-Bernal JM. Fisiopatología de la diabetes y los mecanismos de muerte de las células β pancreáticas. Rev Endocrinol Nutr 2013; 21(3): 98-106.
- [Background] DeFronzo RA, Abdul-Ghani M. Type 2 diabetes can be prevented with early pharmacological intervention. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S202-9. doi: 10.2337/dc11-s221. PMID 21525456
- [Background] D'Adamo E, Caprio S. Type 2 diabetes in youth: epidemiology and pathophysiology. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S161-5. doi: 10.2337/dc11-s212. No abstract available. PMID 21525449
- [Background] Gunawardane K, Krarup Hansen T, Sandahl Christiansen J, Lunde Jorgensen JO Normal physiology of growth hormone in adults. 2015; South Dartmouth, MA: Endotext.
- [Background] Baumann G. Growth hormone binding protein. The soluble growth hormone receptor. Minerva Endocrinol. 2002 Dec;27(4):265-76. PMID 12511849
- [Background] Moller N, Jorgensen JO. Effects of growth hormone on glucose, lipid, and protein metabolism in human subjects. Endocr Rev. 2009 Apr;30(2):152-77. doi: 10.1210/er.2008-0027. Epub 2009 Feb 24. PMID 19240267
- [Background] Krsek M. [Growth hormone, axis GH-IGF1 and glucose metabolism]. Vnitr Lek. 2016 Fall;62(11 Suppl 4):S62-66. Czech. PMID 27921427
- [Background] Goodman y Gilman. Las bases farmacológicas de la terapéutica. 12va. ed. México: McGraw-Hill Interamericana; 2012.
- [Background] Rajpathak SN, Gunter MJ, Wylie-Rosett J, Ho GY, Kaplan RC, Muzumdar R, Rohan TE, Strickler HD. The role of insulin-like growth factor-I and its binding proteins in glucose homeostasis and type 2 diabetes. Diabetes Metab Res Rev. 2009 Jan;25(1):3-12. doi: 10.1002/dmrr.919. PMID 19145587
- [Background] Chang HR, Kim HJ, Xu X, Ferrante AW Jr. Macrophage and adipocyte IGF1 maintain adipose tissue homeostasis during metabolic stresses. Obesity (Silver Spring). 2016 Jan;24(1):172-83. doi: 10.1002/oby.21354. Epub 2015 Dec 10. PMID 26663512
- [Background] Binoux M. The IGF system in metabolism regulation. Diabete Metab. 1995 Dec;21(5):330-7. PMID 8586149
- [Background] Aguirre GA, De Ita JR, de la Garza RG, Castilla-Cortazar I. Insulin-like growth factor-1 deficiency and metabolic syndrome. J Transl Med. 2016 Jan 6;14:3. doi: 10.1186/s12967-015-0762-z. PMID 26733412
- [Background] Clemmons DR. Role of insulin-like growth factor binding proteins in controlling IGF actions. Mol Cell Endocrinol. 1998 May 25;140(1-2):19-24. doi: 10.1016/s0303-7207(98)00024-0. PMID 9722163
- [Background] Hubbard SR, Till JH. Protein tyrosine kinase structure and function. Annu Rev Biochem. 2000;69:373-98. doi: 10.1146/annurev.biochem.69.1.373. PMID 10966463
- [Background] O'Neill BT, Lauritzen HP, Hirshman MF, Smyth G, Goodyear LJ, Kahn CR. Differential Role of Insulin/IGF-1 Receptor Signaling in Muscle Growth and Glucose Homeostasis. Cell Rep. 2015 May 26;11(8):1220-35. doi: 10.1016/j.celrep.2015.04.037. Epub 2015 May 14. PMID 25981038
- [Background] Von Bernhardi M R. Mecanismos de muerte celular en las enfermedades neurodegenerativas: ¿apoptosis o necrosis? Rev Chil Neuro-Psiquiat 2004;42(4):281-92.
- [Background] Navarro M, Baserga R. Limited redundancy of survival signals from the type 1 insulin-like growth factor receptor. Endocrinology. 2001 Mar;142(3):1073-81. doi: 10.1210/endo.142.3.7991. PMID 11181521
- [Background] Miyake H, Kanazawa I, Sugimoto T. Decreased serum insulin-like growth factor-I level is associated with the increased mortality in type 2 diabetes mellitus. Endocr J. 2016 Sep 30;63(9):811-818. doi: 10.1507/endocrj.EJ16-0076. Epub 2016 Jun 25. PMID 27349183
- [Background] Sánchez-Migallón P. Control metabólico en pacientes diabéticos tipo 2: grado de control y nivel de conocimientos (Estudio Azuer) Rev Clin Med Fam 2011; 4(1): 32-4132.
- [Background] Norma Oficial Mexicana NOM-015-SSA2-1994, Para la prevención, tratamiento y control de la diabetes.
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycemia in type 2 diabetes, 2015: a patient-centered approach: update to a position statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2015 Jan;38(1):140-9. doi: 10.2337/dc14-2441. No abstract available. PMID 25538310
- [Background] Panickar K, Cao H, Qin B, Anderson RA. Molecular Targets and Health Benefits of Cinnamon. In: Aggarwal BB, Kunnumakkara AB, editors. Molecular Targets and Therapeutic Uses of Spices. Modern Uses for Ancient Medicine. USA:World Scientific; 2009. p. 87-115.
- [Background] Ziegenfuss TN, Hofheins JE, Mendel RW, Landis J, Anderson RA. Effects of a water-soluble cinnamon extract on body composition and features of the metabolic syndrome in pre-diabetic men and women. J Int Soc Sports Nutr. 2006 Dec 28;3(2):45-53. doi: 10.1186/1550-2783-3-2-45. PMID 18500972
- [Background] Khan A, Safdar M, Ali Khan MM, Khattak KN, Anderson RA. Cinnamon improves glucose and lipids of people with type 2 diabetes. Diabetes Care. 2003 Dec;26(12):3215-8. doi: 10.2337/diacare.26.12.3215. PMID 14633804
- [Background] Blevins SM, Leyva MJ, Brown J, Wright J, Scofield RH, Aston CE. Effect of cinnamon on glucose and lipid levels in non insulin-dependent type 2 diabetes. Diabetes Care. 2007 Sep;30(9):2236-7. doi: 10.2337/dc07-0098. Epub 2007 Jun 11. No abstract available. PMID 17563345
- [Background] Lakshmi BS, Sujatha S, Anand S, Sangeetha KN, Narayanan RB, Katiyar C, Kanaujia A, Duggar R, Singh Y, Srinivas K, Bansal V, Sarin S, Tandon R, Sharma S, Singh S. Cinnamic acid, from the bark of Cinnamomum cassia, regulates glucose transport via activation of GLUT4 on L6 myotubes in a phosphatidylinositol 3-kinase-independent manner. J Diabetes. 2009 Jun;1(2):99-106. doi: 10.1111/j.1753-0407.2009.00022.x. PMID 20929506
- [Background] Ravindran PN, Nirmal Babu K, Shylaja M. Cinnamon and Cassia. The genus Cinnamomum. 2004 CRC Press LLC. Boca Raton Florida, USA.
- [Background] Meena Vangalapati, Sree Satya N, Surya Prakash DV, Sumanjali Avanigadda. A Review on Pharmacological Activities and Clinical effects of Cinnamon Species. RJPBCS 2012; 3(1) 653-663.
- [Background] Nandam Sree Satya, Surya Prakash D.V., Vangalapati Meena. Purification of Cinnamaldehyde from Cinnamon Species by Column Chromatography. Res J Biological Sci 2012: 1(7): 49-51.
- [Background] Jiaju Zhou, Guirong Xie, Xinjian Yan. Encyclopedia of Traditional Chinese Medicines - Molecular Structures, Pharmacological Activities, Natural Sources and Applications: Vol. 4: Isolated Compounds N-S. Editorial Springer-Verlang Berlin Heidelberg 2011. p. 535.
- [Background] Warrier PK, Nambiar VPK, Ramankutty C. Indian Medicinal Plants: A Compendium of 500 Species. Orient Longman, 1994.
- [Background] Cheng DM, Kuhn P, Poulev A, Rojo LE, Lila MA, Raskin I. In vivo and in vitro antidiabetic effects of aqueous cinnamon extract and cinnamon polyphenol-enhanced food matrix. Food Chem. 2012 Dec 15;135(4):2994-3002. doi: 10.1016/j.foodchem.2012.06.117. Epub 2012 Jul 14. PMID 22980902
- [Background] Fugh-Berman A. The 5-minute Herb and Dietary Supplement Consult. Lyppincott Williams & Wilkins 2003. p.86-87.
- [Background] Kirkham S, Akilen R, Sharma S, Tsiami A. The potential of cinnamon to reduce blood glucose levels in patients with type 2 diabetes and insulin resistance. Diabetes Obes Metab. 2009 Dec;11(12):1100-13. doi: 10.1111/j.1463-1326.2009.01094.x. PMID 19930003
- [Background] Kim W, Khil LY, Clark R, Bok SH, Kim EE, Lee S, Jun HS, Yoon JW. Naphthalenemethyl ester derivative of dihydroxyhydrocinnamic acid, a component of cinnamon, increases glucose disposal by enhancing translocation of glucose transporter 4. Diabetologia. 2006 Oct;49(10):2437-48. doi: 10.1007/s00125-006-0373-6. Epub 2006 Aug 9. PMID 16896937
- [Background] Imparl-Radosevich J, Deas S, Polansky MM, Baedke DA, Ingebritsen TS, Anderson RA, Graves DJ. Regulation of PTP-1 and insulin receptor kinase by fractions from cinnamon: implications for cinnamon regulation of insulin signalling. Horm Res. 1998 Sep;50(3):177-82. doi: 10.1159/000023270. PMID 9762007
- [Background] Clemmons DR. Metabolic actions of insulin-like growth factor-I in normal physiology and diabetes. Endocrinol Metab Clin North Am. 2012 Jun;41(2):425-43, vii-viii. doi: 10.1016/j.ecl.2012.04.017. PMID 22682639
- [Background] Jeyaseelan L, Rao PS. Methods of determining sample sizes in clinical trials. Indian Pediatr. 1989 Feb;26(2):115-21. PMID 2753525
- [Background] Brick DJ, Gerweck AV, Meenaghan E, Lawson EA, Misra M, Fazeli P, Johnson W, Klibanski A, Miller KK. Determinants of IGF1 and GH across the weight spectrum: from anorexia nervosa to obesity. Eur J Endocrinol. 2010 Aug;163(2):185-91. doi: 10.1530/EJE-10-0365. Epub 2010 May 25. PMID 20501597
- [Background] Guerrero-Romero F, Simental-Mendia LE, Gonzalez-Ortiz M, Martinez-Abundis E, Ramos-Zavala MG, Hernandez-Gonzalez SO, Jacques-Camarena O, Rodriguez-Moran M. The product of triglycerides and glucose, a simple measure of insulin sensitivity. Comparison with the euglycemic-hyperinsulinemic clamp. J Clin Endocrinol Metab. 2010 Jul;95(7):3347-51. doi: 10.1210/jc.2010-0288. Epub 2010 May 19. PMID 20484475
- [Background] Compendio de Leyes y Reglamentos. Agenda de Salud 2002. Tercera edición. México: Ediciones fiscals ISEF, 2002
- [Background] Surós A, Surós J. Semiología médica y técnica exploratoria. Octava edición. Barcelona: MASSON, 2001
- See also: Pubchem; 2017.Accessed at https://pubchem.ncbi.nlm.nih.gov on 15 June 2017. — http://pubchem.ncbi.nlm.nih.gov